CLINICAL TRIAL: NCT06036056
Title: NMR - Based Metabolomics Approach to Improve Clinical Management in Patients With Respiratory Failure
Brief Title: NMR Based Metabolomics Kinetics in ARDS Patients
Status: Recruiting | Type: Observational
Sponsor: Sanjay Gandhi Postgraduate Institute of Medical Sciences (Other Government)
Collaborators: Centre of BioMedical Research, India (Unknown)
Responsible Party: Principal Investigator, Mohan Gurjar, Professor, Sanjay Gandhi Postgraduate Institute of Medical Sciences
Other Study IDs: 2023-223-CP-133
Record Dates: First submitted 2023-08-31; First posted 2023-09-13 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: ARDS
Keywords: Critically ill; Acute respiratory distress syndrome; Metabolomics; Intensive care unit
MeSH Terms: conditions — Critical Illness; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum of participants will be stored for future research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute Respiratory Distress Syndrome: Mild Acute Respiratory Distress Syndrome
- Healthy: Healthy volunteer

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a life-threatening condition requiring respiratory support to maintain oxygenation. Very few biomarkers about ARDS have been identified but none of them has a sufficient specificity or sensitivity to characterize by itself the severity of lung condition. Investigators hypothesize that there is considerable change occurring in metabolic profiles in mild, moderate, and severe ARDS in comparison to healthy cohort, which can be detectable through serum analysis using NMR based metabolomics study. This research would help to understand metabolomics kinetics during the ARDS disease progression. Overall, NMR-based metabolomics study would provide an insight into the mediators involved in pathogenesis and progression of ARDS.

DETAILED DESCRIPTION:
For this study, all adult ICU patients will be screened for ARDS. Participants who fulfill criteria of mild ARDS (PaO2/FiO2 200-300) will be considered for possible inclusion. For comparative analysis, age matched healthy control will also be included in the study. Investigators are planning to work on the blood samples collected from the participants having mild ARDS. First samples will be collected within 72 hours of fulfilling diagnostic criteria of mild ARDS, thereafter every 72 hours till participants recovered from ARDS or discharge from the ICU or three weeks after inclusion, whichever comes first. For serum preparation, 2 ml of blood samples will be obtained in collection vial, allowed to clot for 60 minutes at room temperature. The samples will then be centrifuged at 1,200 × g for 10 minutes, collected in an eppendorf tubes, sealed and frozen at minus 80 degree Celsius till NMR experiments would be performed. Further 1D and 2D NMR spectroscopic techniques will be used for the characterization and quantitation of various metabolic components of serum.

This study is exploratory in nature to understand kinetics of NMR-based metabolomics in ARDS population. Considering approximately 20-25% of mild ARDS will eventually progress to severe ARDS, investigators will include total 120 participants (including healthy participants). Data collection for comprehends demographic profile, clinical characteristics and illness severity score Sequential Organ Failure Assessment (SOFA) score at the time of study inclusion, clinical course during ICU stay and participants outcome will be done.

NMR spectroscopy (800-MHz Bruker) of sample will be performed using an external tube containing Trimethylsilyl propanoic acid (TSP), D2O to lock the signal. Plasma/Serum samples will be thawed and subsequently centrifuged at 10,000g for 5 min at 4°C to remove any solid debris, 450 μl of each sample will be thoroughly mixed with 50 μl of NMR buffer (1.5 MKH2PO4, 2 mM NaN3, 5.8 mM sodium 3-(trimethylsilyl) propionate-2,2,3,3-d4, D2O, pH 7.4) and the resulting solution will be transferred to 5 mm or 3 mm NMR tubes. All one-dimensional spectra with water suppression will be obtained. Proton spectra will be referenced to the TSP signal (δ=0.00 ppm). The Free induction decays (FIDs) will be processed with line broadening and zero filled before Fourier transformation. The acquired spectra will be manually phased; baseline corrected and integrated using TOPSPIN 2.1.

All NMR spectra will be processed and analysed using TOPSIN 3 package. Auto and supervised peak picking will be performed with Amix and metabolites identification will be done using Metaboanlayst and BIOREFCODE database of metabolites. Standard statistical supervised and unsupervised multivariate analysis (PCA and PLSDA) will be performed.

Metabolites in the 1H NMR spectra of serum samples will be assigned using 1D, 2D, HMDB and BMRB database. Small metabolite overlapping resonances present in 1D spectrum will be confirmed by using 2D spectra including heteronuclear single quantum correlation (HSQC), correlation spectroscopy (COSY), Total correlation spectroscopy (TOCSY), J-resolved (JRES) and Human Metabolome Database and Biological magnetic resonance bank (BMRB) database.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill adult patients having mild ARDS with onset less than 72 hours

Exclusion Criteria:

* Age less than 18 years or more than 65 years
* Expected survival <72 hours
* Refusal from family member

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who fulfill criteria of mild ARDS (PaO2/FiO2 200-300) will be considered for possible inclusion. For comparative analysis, age matched healthy control (from healthy blood donor volunteer will also be included in the study.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-09-13 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
To identify the potential biomarkers in mild ARDS using NMR based metabolomics | Up to the 72 hours after the diagnosis of mild ARDS
  NMR based metabolomics in the serum of patients with mild ARDS
To study the kinetics of NMR based metabolomics in mild ARDS and its association with progression of ARDS severity. | Three weeks after diagnosing mild ARDS or till ICU discharge (whichever comes first)
  Changes in NMR based metabolomics in serum of patients with mild ARDS

SECONDARY OUTCOMES:
Correlation of the infection etiology and NMR based metabolomics | Up to the three weeks after the diagnosis of mild ARDS or ICU discharge (whichever comes first)
  To study microorganism specific changes in NMR based metabolomics, if any

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Sinha, M.Sc., Ph.D., Principal Investigator — Centre of Biomedical Research
Locations (1):
- Centre of Biomedical Research, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Undecided